CLINICAL TRIAL: NCT02775136
Title: An Open-Label, Non-Randomized, Comparative Study Designed to Evaluate the Accuracy and Safety of HS-1000 Device, a Non-Invasive Brain Monitor
Brief Title: An Evaluation of a Non-invasive Brain Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HeadSense Medical (Industry)
Collaborators: Klinikum Stuttgart (Other); Klinikum Darmstadt (Other); University Medical Center Goettingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-011
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2016-12

CONDITIONS: Brain Injuries; Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hydrocephalus; Brain Neoplasms
Keywords: brain injuries; neurological monitoring
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Vasospasm, Intracranial; Hydrocephalus; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): Non-invasive measurements duration with HS-1000 device will be for at least 30 minutes and up to 1 hour of aggregate recording either continuously in the event the patient's clinical condition allows it or in separate recording iterations in the event patient's condition will not allow continuous recording. For each patient, there may be several monitoring intervals from three times a day and up to as long as the patient undergoes brain monitoring, per the discretion of the investigator, patient and/or family members.
  Interventions: Device: HS-1000 recording

INTERVENTIONS:
Device: HS-1000 recording

SUMMARY:
HS-1000 device, a proprietary new non-invasive brain monitor, is expected to safely and accurately monitor physiological signs of the brain with minimal discomfort to patients, providing information about normal or abnormal brain-related conditions and providing decision-making support for physicians. Investigators hypothesis that the HS-1000 is capable of detecting and monitoring various neuropathologies, using the acoustic raw data derived from the noninvasive procedure.

DETAILED DESCRIPTION:
Non-invasive modality for brain monitoring can potentially serve as a major contribution to conventional monitoring techniques for patients with neuropathologies, to assure minimal discomfort to the bedbound patients, and provide information about critical physiological signs to the physicians. The lack of a precise diagnostic technique for numerous neuropathologies for patients in neurosurgical clinics can further hinder therapeutic effectiveness and, therefore, influence patient recovery and healing. Neuro-critical care involves monitoring standard vital signs and cerebral physiological signs, mainly focusing on intracranial pressure (ICP), temperature, cerebral blood flow velocity, arterial blood pressure, cerebral perfusion pressure, brain tissue oxygenation etc. The collaboration of state of the art brain monitoring vary between different intensive care units serves a significant drawback in some cases, as accuracy of diagnosis and monitoring is challenged and thereby there is an eminent need for interrelationship brain monitoring approach. That can also be leveraged by applying the monitoring noninvasively, as it particularly beneficial for clinical applications that routinely require the inevitable and dynamic transport of patients between hospital units (imaging, surgical room, etc.).

Subjects who meet the inclusion and exclusion criteria for this study, with a signed informed consent form, will be enrolled into the study. Eligible patients will be divided to 2 groups:

1. Patients undergoing Invasive ICP monitoring
2. Subarachnoid hemorrhage (SAH) patients with Fisher Grade of 3 or 4

The non-invasive measurements recording sessions will be according to the protocol scheme per each group:

1. Eligible patients undergoing Invasive ICP monitoring will be monitored by the HS-1000, in parallel to the invasive ICP monitor, for a single recording session.
2. Eligible SAH patients with Fisher Grade of 3 or 4 will be monitored by the HS-1000, in parallel to the invasive ICP monitor, for three recording sessions.

For all eligible patients, non-invasive measurements by the HS-1000 device will be conducted in parallel with the standard monitoring modalities, as used at the site without any change in the patient's management.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women subjects, aged 18 years old and over at screening visit
2. Subjects with neuropathology that the principal investigator considers including in this study.
3. Survival expectancy greater than 72 hours
4. Subject or legal authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
5. Subject or legal authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

1. Local ear infection
2. Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
3. For women of childbearing potential: pregnancy (positive pregnancy test) or breast-feeding
4. Subarachnoid hemorrhage (SAH), Fisher Grade 4
5. Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
6. Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of recordings that correlate to neuropathology | up to 1 hour
  Demonstrate the HS-1000 performance and accuracy in brain monitoring

SECONDARY OUTCOMES:
Incidence of adverse events | 48 hours from the end of monitoring with the HS-1000
Rate of ear infections/irritations graded by none/mild/moderate and severe | 48 hours from the end of monitoring with the HS-1000

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Ganslandt, Prof., Principal Investigator — Klinikum Stuttgart
Locations (4):
- Germany (4):
  - Klinikum Darmstadt, Darmstadt
  - University Hospital Erlangen, Erlangen
  - Universitätsklinik Göttingen, Göttingen
  - Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No